CLINICAL TRIAL: NCT02814578
Title: Assessment of Coronary Artery Lesion Using Optical Coherence Tomography Versus IntraVascular Ultrasound for BiorEsorbable Vascular Scaffold Implantation
Acronym: ACTIV-BVS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: OCT cost is high
Sponsor: Young-Hak Kim, MD, PhD (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, Young-Hak Kim, MD, PhD, Professor in medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMCCV2016-02
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
Keywords: OCT; IVUS; BVS
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optical coherent tomography (Experimental): Optical coherent tomography provides more detailed information about the morphology of scaffolds, microstructures and coronary vasculature based on tissue characteristics as compared to conventional IVUS. In spite of angiographic success in BVS placement, further scaffold optimization was required in over a quarter of cases based on OCT findings due to malapposition or scaffold under expansion.
  Interventions: Other: Optical coherent tomography
- IntraVascular UltraSound (Active Comparator): Intravascular ultrasound guidance has been associated with improved event-free survival compared with angiographic guidance after DES placement.
  Interventions: Other: IntraVascular UltraSound

INTERVENTIONS:
Other: Optical coherent tomography — comparative method for BVS
  Arms: Optical coherent tomography
Other: IntraVascular UltraSound — The method of goldstandard for decision stent choice
  Arms: IntraVascular UltraSound

SUMMARY:
The primary objective is to determine whether IVUS- (vs. OCT-) guided BVS implantation is non-inferior to achieve a large in-scaffold minimal lumen area (primary endpoint) measured by OCT at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older
* Patients who have at least one epicardial coronary artery lesion with an evidence of inducible ischemia
* Willing and able to provide informed written consent
* Eligible for PCI

Exclusion Criteria:

* Patients presenting with STEMI within 2 weeks
* Bypass graft lesion
* Lesion with left main disease
* Expected length of scaffold > 40 mm
* Bifurcation lesion requiring side branch stenting
* Small vessels < 2.75 mm
* Stented lesion
* Suspected coronary spasm even after sufficient nitrate injected
* Cases in which the IVUS or OCT imaging catheter failed to cross the lesion
* Poor quality IVUS or OCT images
* Contraindication to dual anti-platelet therapy
* Chronic total occlusion
* Angiographically large-sized vessel (>3.5mm of reference lumen diameter)
* Life expectancy shorter than 2 years
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
OCT-measured in-scaffold minimal lumen area | 1 year

SECONDARY OUTCOMES:
OCT-measured minimal scaffold area (MSA) | 1 year
OCT-measured mean scaffold expansion | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul, Songpa-Gu
  - Pusan National University Hospital, Pusan
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.